CLINICAL TRIAL: NCT00207766
Title: ACCENT II - A Randomized, Double-blind, Placebo-controlled Trial of Anti-TNF Chimeric Monoclonal Antibody (Infliximab, Remicade) in the Long Term Treatment of Patients With Fistulizing CROHN'S Disease
Brief Title: A Study of the Safety and Efficacy of Infliximab (Remicade) in Subjects With Fistulizing Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005413
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2009-01

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; infusions
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

INTERVENTIONS:
Drug: infliximab or placebo

SUMMARY:
A study of infliximab in patients with Fistulizing Crohn's Disease

DETAILED DESCRIPTION:
This is a medical research study for patients with Crohn's disease who have one or more draining enterocutaneous fistula (fistula from the bowel to the skin). Fistulas are a common complication of Crohn's disease. Fistulas rarely close spontaneously but they may get better with treatment of the underlying Crohn's disease. This study will investigate the safety and efficacy of maintenance dosing of an anti-TNF (anti-tumor necrosis factor) antibody (a protein), called infliximab, compared to a placebo (inactive substance) in providing sustained reductions in the number of draining fistulas.

Subjects will receive infliximab at weeks 0, 2 and 6 followed by infusions of infliximab 5 mg/kg or placebo at weeks 14 and every 8 weeks until week 46. Patients who lose response are eligible for increasing treatment by 5 mg/kg of infliximab.

ELIGIBILITY:
Inclusion Criteria:

* Single or multiple draining fistulas
* Crohn's disease of at least 3 months' duration,

Exclusion Criteria:

* Crohn's disease complications for which surgery might be indicated
* Positive stool culture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2000-06; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Reduction in the number of draining fistulas

SECONDARY OUTCOMES:
Complete fistula response (no draining fistula).

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Sands BE, Blank MA, Patel K, van Deventer SJ; ACCENT II Study. Long-term treatment of rectovaginal fistulas in Crohn's disease: response to infliximab in the ACCENT II Study. Clin Gastroenterol Hepatol. 2004 Oct;2(10):912-20. doi: 10.1016/s1542-3565(04)00414-8. PMID 15476155
- [Result] Sands BE, Anderson FH, Bernstein CN, Chey WY, Feagan BG, Fedorak RN, Kamm MA, Korzenik JR, Lashner BA, Onken JE, Rachmilewitz D, Rutgeerts P, Wild G, Wolf DC, Marsters PA, Travers SB, Blank MA, van Deventer SJ. Infliximab maintenance therapy for fistulizing Crohn's disease. N Engl J Med. 2004 Feb 26;350(9):876-85. doi: 10.1056/NEJMoa030815. PMID 14985485